CLINICAL TRIAL: NCT00545363
Title: A Randomized Open-Label Study to Investigate the Impact of Bone Marker Feedback at 3 Months on Adherence to Monthly Oral Bonviva in Women With Post-Menopausal Osteoporosis Supported by a Patient Relationship Program
Brief Title: A Study of Adherence to Once Monthly Ibandronate (Bonviva) in Women With Post-Menopausal Osteoporosis, Supported by a Patient Relationship Program (PRP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19982; 2005-005529-74 (EudraCT Number)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (2):
- Bone Marker Feedback (BMF) Participants (Experimental): Postmenopausal women will receive ibandronate 150 milligrams (mg) once monthly (QM) orally for 6 months. Participants, in this arm, will receive BMF at Month 3. BMF will be given in terms of providing serum carboxy-terminal collagen crosslinks (CTX) level at Month 3. A "BMF-form" will be provided to the physicians to allow offering the bone marker result in an easy way. Participants will be informed if their results are within or outside of the desired range. In addition, participants will also supported by PRP, to be carried out by supplying alarm devices, specifically designed to support the participant's regular drug intake.
  Interventions: Drug: Ibandronate
- No BMF Participants (Active Comparator): Postmenopausal women will receive ibandronate 150 milligrams (mg) once monthly (QM) orally for 6 months. Participants will be supported by PRP, to be carried out by supplying alarm devices, specifically designed to support the participant's regular drug intake.
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Participants will receive ibandronate 150 mg QM orally for 6 months.
  Other Names: Bonviva; Boniva

SUMMARY:
This 2 arm study will assess the impact of bone marker feedback (BMF), using serum carboxy-terminal collagen crosslinks (CTX) and communication of results at 3 months, on adherence to once monthly ibandronate (150 milligrams [mg] per oral [po]) in women with post-menopausal osteoporosis supported by patient-relationship program (PRP). Participants will be randomized either to receive BMF or no BMF; both groups will be supported by PRP. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory, post-menopausal women with osteoporosis;
* eligible for bisphosphonate treatment;
* naïve to bisphosphonate therapy, or lapsed users (last bisphosphonate intake greater than or equal to [>=] 6 months ago).

Exclusion Criteria:

* inability to stand or sit upright for at least 60 minutes;
* inability to swallow a tablet whole;
* hypersensitivity to bisphosphonates;
* treatment with drugs, or presence of active disease, known to influence bone metabolism;
* history of upper gastrointestinal disease.

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Hungary (8):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Miskolc
  - Pécs
  - Szeged
  - Székesfehérvár
  - Szombathely
- Latvia (2):
  - Liepāja
  - Riga
- Poland (6):
  - Gliwice
  - Krakow
  - Lodz
  - Poznan
  - Warsaw
  - Wroclaw
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Craiova
  - Timișoara
- Russia (6):
  - Irkutsk
  - Moscow
  - Saint Petersburg
  - Voronezh
  - Yaroslavl
  - Yekaterinburg
- Slovakia (5):
  - Banská Bystrica
  - Bratislava
  - Ľubochňa
  - Piešťany
  - Prešov
- Ljubljana, Slovenia

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marker Feedback (BMF) Participants: Postmenopausal women received ibandronate 150 milligrams (mg) once monthly (QM) orally for 6 months. Participants, in this arm, received bone marker feedback (BMF) at Month 3. BMF was given in terms of providing serum carboxy-terminal collagen crosslinks (CTX) level at Month 3. A "BMF-form" was provided to the physicians to allow offering the bone marker result in an easy way. Participants were informed that their results were within or outside of the desired range. In addition, participants were also supported by patient relationship program (PRP), carried out by supplying alarm devices, specifically designed to support the participant's regular drug intake.
- No BMF Participants: Postmenopausal women received ibandronate 150 mg QM orally for 6 months. Participants were supported by PRP, carried out by supplying alarm devices, specifically designed to support the participant's regular drug intake.
Period: Overall Study
Arm/Group | Bone Marker Feedback (BMF) Participants | No BMF Participants
Started | 358 | 358
Treated | 354 | 357
Completed | 339 | 343
Not Completed | 19 | 15
Not completed — Adverse Event | 6 | 7
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Non-compliance | 3 | 1
Not completed — Did not meet entry criteria | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received at least 1 dose of study drug.
Groups:
- BMF Participants: Postmenopausal women received ibandronate 150 mg QM orally for 6 months. Participants, in this arm, received BMF at Month 3. BMF was given in terms of providing serum CTX level at Month 3. A "BMF-form" was provided to the physicians to allow offering the bone marker result in an easy way. Participants were informed that their results were within or outside of the desired range. In addition, participants were also supported by PRP, carried out by supplying alarm devices, specifically designed to support the participant's regular drug intake.
- Total: Total of all reporting groups
Arm/Group | BMF Participants | No BMF Participants | Total
Number analyzed (Participants) | 354 | 357 | 711
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (7.12) | 65.6 (6.64) | 66.2 (6.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 354 | 357 | 711
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adherence to Treatment
Description: Participants were considered adherent to treatment if they took at least 83 percent (%) of their assigned medications (5 of the 6 monthly ibandronate tablets) within the -1 to +21 days of their osteoporosis treatment date each month. Participant adherence was assessed by maintaining records of 'drug dispensed' and 'drug returned' on case report form (CRF) and participant's self-report on Visit 2 (Month 3) and final study visit (Month 6). A drug dispensing log was maintained by the investigator. Participants were instructed at the baseline visit and Visit 2 to save and return unused or partially used medication packages on Visit 2 and final study visit, respectively.
Time Frame: Up to 6 months
Population: Intent to treat (ITT) population included all randomized participants. Number of participants analyzed=number of participants evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | BMF Participants | No BMF Participants
Number analyzed (Participants) | 271 | 284
percentage of participants | 98.5 | 98.6

2. Secondary Outcome: Percentage of Participants With Osteoporosis Patient Satisfaction Questionnaire (OPSAT-Q) Composite Satisfaction High Scores
Description: The OPSAT-Q is a validated questionnaire designed to capture satisfaction with bisphosphonate treatment. It comprises four domains: convenience (questions 1 - 6), quality of life (questions 7 and 8), overall satisfaction (questions 9 and 10), and side effects (questions 11 - 16). Satisfaction with treatment was assessed using the OPSAT-Q composite satisfaction score, which was the average of the scores from the four domains of the OPSAT-Q converted to a 0 - 100-point scale. Higher scores indicated greater treatment satisfaction. A score of 80 or more was considered as high score.
Time Frame: At Month 6
Population: ITT population. Number of participants analyzed = participants evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | BMF Participants | No BMF Participants
Number analyzed (Participants) | 328 | 336
percentage of participants | 87.72 | 87.62
Statistical Analysis 1: Comparison: BMF Participants vs No BMF Participants; Statistical analysis was done to compare the participant satisfaction between the Biofeedback and No-feedback arms; Test type: Superiority or Other; p = 0.8989, ANOVA

3. Secondary Outcome: Percentage of Participants With Osteoporosis Patient Perception Survey (OPPS) and Osteoporosis Medical Care Satisfaction Questionnaire (OMSQ) Composite Satisfaction High Score
Description: OPPS: A standardized 6-item satisfaction questionnaire for osteoporosis medical care and treatment received during the study. Individual item score was transformed and converted to a 0 to 100 scale where higher score indicated greater satisfaction. The composite score was the average of individual item scores (transformed) and ranged from 0 to 100, where higher scores indicated greater satisfaction. OMSQ: A standardized 18-item satisfaction questionnaire for osteoporosis medical care, treatment received and blood test and their results during the study. Individual item score was transformed and converted to a 0 to 100 scale where higher score indicated greater satisfaction. The composite score was the average of individual item scores (transformed) and ranged from 0 to 100, where higher scores indicated greater satisfaction.
Time Frame: At Month 6
Population: ITT population. Number of participants analyzed = participants evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | BMF Participants | No BMF Participants
Number analyzed (Participants) | 328 | 334
percentage of participants | 74.9 | 72.2
Statistical Analysis 1: Comparison: BMF Participants vs No BMF Participants; Statistical analysis was done to compare the participant perception between the Biofeedback and No-feedback arms; Test type: Superiority or Other; p = 0.453, ANOVA

4. Secondary Outcome: Percent Change From Baseline in CTX Based on Adherence to Ibandronate
Description: Serum CTX, a biochemical marker of bone resorption, was assessed for all participants at baseline and at final visit (Month 6). The sampling was done at the same time of the day each time to overcome the effect of circadian fluctuations. Participants were considered adherent to treatment if they took at least 83% of their assigned medications (5 of the 6 monthly ibandronate tablets) within the -1 to +21 days of their osteoporosis treatment date each month. Participant adherence was assessed by maintaining records of 'drug dispensed' and 'drug returned' on CRF and participant's self-report on Visit 2 (Month 3) and final study visit (Month 6). A drug dispensing log was maintained by the investigator. Participants were instructed at the baseline visit and Visit 2 to save and return unused or partially used medication packages on Visit 2 and final study visit, respectively.
Time Frame: Baseline, Month 6
Population: ITT population. Number of participants analyzed = participants evaluable for this outcome and "n" represents number of participants analyzed for the specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | BMF Participants | No BMF Participants
Number analyzed (Participants) | 280 | 287
percent change
  Adherence-Yes (n=279, 281) | -47.5 [-51.3 to -43.5] | -47.5 [-51.0 to -43.9]
  Adherence-No (n=1, 6) | -71.74 [NA to NA] — Standard deviation is not applicable as there is only 1 participant. | -25.8 [-91.0 to 13.5]
Statistical Analysis 1: Comparison: BMF Participants vs No BMF Participants; Statistical analysis was done to compare the effect of adherence (Yes/No) on percent change from baseline in CTX between the Biofeedback and No-feedback arms; Test type: Superiority or Other; p = 0.4917, ANOVA

ADVERSE EVENTS:
Time Frame: 15-30 days after final visit (final visit=up to 6 months)
Arm/Group | BMF Participants | No BMF Participants
Serious Adverse Events (participants affected / at risk) | 8/354 | 5/357
Other Adverse Events (participants affected / at risk) | 196/354 | 224/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMF Participants (N=354) | No BMF Participants (N=357)
Cardiac arrest (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMF Participants (N=354) | No BMF Participants (N=357)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 0
Tricuspid valve disease (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Cataract (Eye disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Keratopathy (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Abdominal pain upper (Gastrointestinal disorders) | 5 | 9
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 12
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 10
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Glossitis (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 10 | 5
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Acute phase reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Hyperthermia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 4 | 1
Malaise (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 2
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 5
Cellulitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 5 | 3
Fungal infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 3 | 4
Nasopharyngitis (Infections and infestations) | 6 | 10
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 3 | 4
Pneumonia (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 6 | 4
Viral infection (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Burn oesophageal (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Near drowning (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose increased (Investigations) | 2 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Laboratory test abnormal (Investigations) | 1 | 0
Urine output increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Lipid metabolism disorder (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 4 | 7
Migraine (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Panic disorder (Psychiatric disorders) | 1 | 1
Calculus urinary (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Glaucoma surgery (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 1
Arteriosclerosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 4 | 4
Labile blood pressure (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.